CLINICAL TRIAL: NCT01737996
Title: An Open-label, Multiple Dose Study to Assess Safety, Tolerability and Pharmacokinetics of Different Multiple Doses of BI 207127 BID Administered Orally for 9 Days (Part 1) and Multiple Doses of BI 207127 Combined With Faldaprevir Administered Orally for 16 Days (Part 2) in Healthy Male and Female Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Different Multiple Doses of BI 207127 BID and Multiple Doses of BI 207127 Combined With Faldaprevir in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1241.35; 2012-003697-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-11-26; First posted 2012-11-30 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — deleobuvir; faldaprevir

ARMS (1):
- All patients (Experimental): For the first 9 days patients receive BI 207127 low dose or high dose, then BI 207127 high dose with faldaprevir
  Interventions: Drug: BI 207127 + faldaprevir

INTERVENTIONS:
Drug: BI 207127 + faldaprevir — fixed dose combination

SUMMARY:
The objective of the current trial is to evaluate safety, tolerability and pharmacokinetics of different multiple doses of BI 207127 BID and multiple doses of BI 207127 combined with faldaprevir in healthy male and female subjects.

ELIGIBILITY:
Inclusion criteria:

1. healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.35.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 600mg dose cohort was to be started at least 6 days after the 400mg dose cohort was completed and the combined treatment cohort (600mg Deleobuvir + 120mg Faldaprevir) was started after the evaluation of key safety and tolerability data of the individual treatments.
Groups:
- 400 mg Deleobuvir: 400 mg Deleobuvir administered twice daily for 9 days. Oral administration with 240 mL of water under fed conditions. Low dose of multiple rising dose (MRD) part.
- 600 mg Deleobuvir: 600 mg Deleobuvir administered twice daily for 9 days. Oral administration with 240 mL of water under fed conditions. Low dose of multiple rising dose (MRD) part.
- 600 mg Deleobuvir + 120 mg Faldaprevir: 600 mg Deleobuvir administered twice daily and 120 mg Faldaprevir administered once daily for 16 days.
  Oral administration with 240 mL of water under fed conditions. Combined treatment part; conducted after multiple rising dose part.
Period: Overall Study
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir | 600 mg Deleobuvir + 120 mg Faldaprevir
Started | 8 | 8 | 16
Completed | 8 | 7 | 14 (One patient withdrew consent after the first dose due to private reasons.)
Not Completed | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study comprised 2 trial parts: a multiple rising dose part (Part 1) followed by a combined treatment part (Part 2). The multiple rising dose part was performed in an open-label, non-randomised, non-placebocontrolled manner with 2 dose groups. The combined treatment part was conducted open-label in 1 treatment group.
Groups:
- 400 mg Deleobuvir: 400 mg Deleobuvir administered twice daily for 9 days. Oral administration with 240 mL of water under fed conditions. Low dose of multiple rising dose part.
- 600 mg Deleobuvir: 600 mg Deleobuvir administered twice daily for 9 days. Oral administration with 240 mL of water under fed conditions. High dose of multiple rising dose part.
- Total: Total of all reporting groups
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir | 600 mg Deleobuvir + 120 mg Faldaprevir | Total
Number analyzed (Participants) | 8 | 8 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.4) | 37.3 (5.1) | 38.3 (10.6) | 38.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 6 | 13
  Male | 5 | 4 | 10 | 19

OUTCOME MEASURES:

1. Secondary Outcome: AUC(0-12h) and AUC(0-12h,ss) of Deleobuvir (Multiple Rising Dose Part)
Description: Area under the concentration-time curve of Deleobuvir over the uniform dosing interval 0 to 12 h on Day 1 and at steady state on Day 9.
Time Frame: After the first administration of Deleobuvir on Day 1 and after the last administration on Day 9: at 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8,12 h after drug administration in the morning.
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 7
nmol*h/L
  AUC(0-12h) on Day 1 | 8210 (45.5) | 18000 (77.6)
  AUC(0-12h,ss) on Day 9 | 6160 (45.2) | 18500 (93.3)

2. Primary Outcome: Number of Healthy Subjects With AEs (Multiple Rising Dose Part)
Description: Number of healthy subjects with any adverse event (AE) during the on-treatment period.
Time Frame: From first drug administration (Day 1) until end of trial examination (15 to 21 days after first administration)
Population: Treated Set. The treated set included all subjects who were documented to have taken at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 8
participants | 6 | 5

3. Primary Outcome: AUC(0-12h) and AUC(0-12h,ss) of Deleobuvir (Combined Treatment Part)
Description: Area under the concentration-time curve (AUC) of Deleobuvir over the uniform dosing interval 0 to 12 h (hours) on Day 1 and at steady state on Day 16.
Time Frame: After the first administration of Deleobuvir+Faldaprevir on Day 1 and after the last administration on Day 16 at 0 (5 min before administration on Day 16), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8,12 hours (h) after drug administration in the morning.
Population: PKS. The pharmacokinetic set (PKS) included all subjects of the treated set who provided at least 1 observation for at least 1 pharmacokinetic endpoint without important protocol violations relevant for the statistical evaluation of pharmacokinetic endpoints. Including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol*h/L
  AUC(0-12h) on Day 1 | 37500 (49.4)
  AUC(0-12h,ss) on Day 16 | 51400 (57.2)

4. Primary Outcome: Cmax and Cmax,ss of Deleobuvir (Combined Treatment Part)
Description: Maximum measured concentration of Deleobuvir on Day 1 and at steady state on Day 16.
Time Frame: After the first administration of Deleobuvir+Faldaprevir on Day 1 and after the last administration on Day 16 at 0 (5 min before administration on Day 16), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8,12 h after drug administration in the morning.
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 15
nmol/L
  Cmax on Day 1 | 6930 (47.9)
  Cmax,ss on Day 16 (N=14) | 9710 (43.3)

5. Primary Outcome: C(12h) and C(12h,ss) of Deleobuvir (Combined Treatment Part)
Description: Concentration of Deleobuvir at the end of the dosing interval 0 to 12 h on Day 1 and at steady state on Day 16.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol/L
  C(12h) on Day 1 | 1090 (69.3)
  C(12h,ss) on Day 16 | 1000 (85.9)

6. Primary Outcome: AUC(0-12h) and AUC(0-12h,ss) of CD 6168 (Combined Treatment Part)
Description: Area under the concentration-time curve of CD 6168 over the uniform dosing interval 0 to 12 h on Day 1 and at steady state on Day 16.
  CD 6168 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol*h/L
  AUC(0-12h) on Day 1 | 6080 (55.0)
  AUC(0-12h,ss) on Day 16 | 38100 (76.0)

7. Secondary Outcome: Cmax and Cmax,ss of Deleobuvir (Multiple Rising Dose Part)
Description: Maximum measured concentration of Deleobuvir on Day 1 and at steady state on Day 9.
Time Frame: as for outcome 1
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 7
nmol/L
  Cmax on Day 1 | 2010 (41.5) | 3740 (79.4)
  Cmax,ss on Day 9 | 1380 (48.3) | 3650 (91.6)

8. Secondary Outcome: AUC(0-12h) and AUC(0-12h,ss) of CD 6168 (Multiple Rising Dose Part)
Description: Area under the concentration-time curve of CD 6168 over the uniform dosing interval 0 to 12 h on Day 1 and at steady state on Day 9.
  CD 6168 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 1
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 7
nmol*h/L
  AUC(0-12h) on Day 1 | 1690 (56.0) | 2920 (88.3)
  AUC(0-12h,ss) on Day 9 | 2810 (63.1) | 6960 (106.0)

9. Secondary Outcome: Cmax and Cmax,ss of CD 6168 (Multiple Rising Dose Part)
Description: Maximum measured concentration of CD 6168 on Day 1 and at steady state on Day 9.
  CD 6168 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 1
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 7
nmol/L
  Cmax on Day 1 | 329 (60.5) | 516 (92.7)
  Cmax,ss on Day 9 | 451 (66.3) | 1130 (90.9)

10. Secondary Outcome: AUC(0-12h) and AUC(0-12h,ss) of BI 208333 (Multiple Rising Dose Part)
Description: Area under the concentration-time curve of BI 208333 over the uniform dosing interval 0 to 12 h on Day 1 and at steady state on Day 9.
  BI 208333 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 1
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 7
nmol*h/L
  AUC(0-12h) on Day 1 | 3940 (38.7) | 6060 (57.1)
  AUC(0-12h,ss) on Day 9 | 2840 (51.7) | 5270 (102.0)

11. Secondary Outcome: Cmax and Cmax,ss of BI 208333 (Multiple Rising Dose Part)
Description: Maximum measured concentration of BI 208333 on Day 1 and at steady state on Day 9.
  BI 208333 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 1
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 7
nmol/L
  Cmax on Day 1 | 766 (41.5) | 1050 (54.2)
  Cmax,ss on Day 9 | 576 (44.4) | 983 (82.4)

12. Secondary Outcome: AUC(0-12h) and AUC(0-12h,ss) of CD 6168 Acylglucuronide (Multiple Rising Dose Part)
Description: Area under the concentration-time curve of CD 6168 acylglucuronide over the uniform dosing interval 0 to 12 h on Day 1 and at steady state on Day 9.
  CD 6168 acylglucuronide is a metabolite of Deleobuvir.
Time Frame: as for outcome 1
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 7 | 7
nmol*h/L
  AUC(0-12h) on Day 1 | 155 (27.2) | 342 (66.0)
  AUC(0-12h,ss) on Day 9 (N=6, 7) | 256 (42.7) | 701 (94.0)

13. Secondary Outcome: Cmax and Cmax,ss of CD 6168 Acylglucuronide (Multiple Rising Dose Part)
Description: Maximum measured concentration of CD 6168 acylglucuronide on Day 1 and at steady state on Day 9.
  CD 6168 acylglucuronide is a metabolite of Deleobuvir.
Time Frame: as for outcome 1
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir
Number analyzed (Participants) | 8 | 7
nmol/L
  Cmax on Day 1 | 27.3 (36.8) | 57.9 (61.0)
  Cmax,ss on Day 9 | 33.3 (61.3) | 116.0 (80.6)

14. Primary Outcome: Cmax and Cmax,ss of CD 6168 (Combined Treatment Part)
Description: Maximum measured concentration of CD 6168 on Day 1 and at steady state on Day 16.
  CD 6168 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol/L
  Cmax on Day 1 | 902 (49.2)
  Cmax,ss on Day 16 | 4860 (60.5)

15. Primary Outcome: C(12h) and C(12h,ss) of CD 6168 (Combined Treatment Part)
Description: Concentration of CD 6168 at the end of the dosing interval 0 to 12 h on Day 1 and at steady state on Day 16.
  CD 6168 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol/L
  C(12h) on Day 1 | 488 (67.5)
  C(12h,ss) on Day 16 | 1650 (102.0)

16. Primary Outcome: AUC(0-12h) and AUC(0-12h,ss) of BI 208333 (Combined Treatment Part)
Description: Area under the concentration-time curve of BI 208333 over the uniform dosing interval 0 to 12 h on Day 1 and at steady state on Day 16.
  BI 208333 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol*h/L
  AUC(0-12h) on Day 1 | 9130 (46.9)
  AUC(0-12h,ss) on Day 16 | 13600 (71.1)

17. Primary Outcome: Cmax and Cmax,ss of BI 208333 (Combined Treatment Part)
Description: Maximum measured concentration of BI 208333 on Day 1 and at steady state on Day 16.
  BI 208333 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 15
nmol/L
  Cmax on Day 1 | 1450 (40.0)
  Cmax,ss on Day 16 (N=14) | 2060 (57.6)

18. Primary Outcome: C(12h) and C(12h,ss) of BI 208333 (Combined Treatment Part)
Description: Concentration of BI 208333 at the end of the dosing interval 0 to 12 h on Day 1 and at steady state on Day 16.
  BI 208333 is a major metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol/L
  C(12h) on Day 1 | 520 (80.8)
  C(12h,ss) on Day 16 | 447 (101.0)

19. Primary Outcome: AUC(0-12h) and AUC(0-12h,ss) of CD 6168 Acylglucuronide (Combined Treatment Part)
Description: Area under the concentration-time curve of CD 6168 acylglucuronide over the uniform dosing interval 0 to 12 h on Day 1 and at steady state on Day 16.
  CD 6168 acylglucuronide is a metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol*h/L
  AUC(0-12h) on Day 1 | 511 (69.9)
  AUC(0-12h,ss) on Day 16 | 3560 (120.0)

20. Primary Outcome: Cmax and Cmax,ss of CD 6168 Acylglucuronide (Combined Treatment Part)
Description: Maximum measured concentration of CD 6168 acylglucuronide on Day 1 and at steady state on Day 16.
  CD 6168 acylglucuronide is a metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 15
nmol/L
  Cmax on Day 1 | 83.9 (63.7)
  Cmax,ss on Day 16 (N=14) | 457.0 (106.0)

21. Primary Outcome: C(12h) and C(12h,ss) of CD 6168 Acylglucuronide (Combined Treatment Part)
Description: Concentration of CD 6168 acylglucuronide at the end of the dosing interval 0 to 12 h on Day 1 and at steady state on Day 16.
  CD 6168 acylglucuronide is a metabolite of Deleobuvir.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol/L
  C(12h) on Day 1 | 56.4 (67.1)
  C(12h,ss) on Day 16 | 178.0 (122.0)

22. Primary Outcome: AUC(0-24h) and AUC(0-24h,ss) of Faldaprevir (Combined Treatment Part)
Description: Area under the concentration-time curve of Faldaprevir over the uniform dosing interval 0 to 24 h on Day 1 and at steady state on Day 16.
Time Frame: as for outcome 4
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 14
nmol*h/L
  AUC(0-12h) on Day 1 | 44800 (23.6)
  AUC(0-12h,ss) on Day 16 | 66200 (46.1)

23. Primary Outcome: Cmax and Cmax,ss of Faldaprevir (Combined Treatment Part)
Description: Maximum measured concentration of Faldaprevir on Day 1 and at steady state on Day 16.
Time Frame: After the first administration of Deleobuvir+Faldaprevir on Day 1 and after the last administration on Day 16 at 0 (5 min before administration on Day 16), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8,12, 24 h after drug administration in the morning.
Population: PKS including patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600 mg Deleobuvir + 120 mg Faldaprevir
Number analyzed (Participants) | 15
nmol/L
  Cmax on Day 1 | 4060.0 (25.0)
  Cmax,ss on Day 16 (N=14) | 5940.0 (32.3)

ADVERSE EVENTS:
Time Frame: From first drug administration (Day 1) until end of trial examination (15 to 21 days after first administration)
Description: Subjects were required to report spontaneously any AEs. In addition, each subject was assessed by the investigator at pre-defined timepoints and whenever it was deemed necessary by the investigator.
Arm/Group | 400 mg Deleobuvir | 600 mg Deleobuvir | 600 mg Deleobuvir + 120 mg Faldaprevir
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 6/8 | 5/8 | 9/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 400 mg Deleobuvir (N=8) | 600 mg Deleobuvir (N=8) | 600 mg Deleobuvir + 120 mg Faldaprevir (N=16)
Folliculitis (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 5
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2
Transaminases increased (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.